CLINICAL TRIAL: NCT06114316
Title: Effect of Interventions Based on Roy Adaptation Model on the Recovery of Individuals With Alcohol Use Disorders: A Randomized Trial
Brief Title: Recovery of Individuals With Alcohol Use Disorders Based on Roy Adaptation Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Dilek AYAKDAS DAGLI, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ayakdasdaglı
Record Dates: First submitted 2023-10-02; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Addiction, Alcohol
Keywords: recovery; alcohol use disorder; Roy Adapation model; Nursing Intervention
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Eighty individuals who alcohol use disorder were assessed for eligibility and 70 individuals (who completed their detoxification process, were able to understand the scales and forms and maintain individual interviews, were between 30 and 60 years of age, were diagnosed with alcohol addiction according to the DSM-5 diagnostic criteria, and voluntarily agreed to participate in the studywere) randomized. An experimental and a control group were formed by assigning persons to each group by using the stratified randomization technique in which a sex factor was involved, according to a random-number table. Four male participants in the experimental group (who were not involved in intervention) and two male participants in the control group (who were discharged) were excluded as they did not continue the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): The control group continued to receive routine treatment (pharmacotherapy and psychoeducation) and follow-up in the Alcohol and Substance Addiction Treatment Center, and no intervention was made.
- experimental (Active Comparator): In the first step, the stimuli that led the individuals in the experimental group to drink alcohol were assessed, and the conceptual-theoretical-experimental (CTE) framework of the study was created. The personal behaviors that could be related to recurrence (physiological, self-concept, role function, and mutual commitment) and the stimuli that caused recurrence (focal and affecting) were assessed, objectives were determined, and nursing interventions were carried out in line with these objectives. The interventions planned for diagnosing ineffective coping were selected according to the patients' needs among the "support coping" interventions under the title of the behavioral area in the Nursing Intervention Classification (NIC). A total of 10 individual interviews were made twice a week for about 45 to 60 minutes. The interviews were evaluated by determining the area specific Nursing outcome classification (NOC) (self respect, social support, mood management, role performance).
  Interventions: Behavioral: individualized nursing interventions based on the Roy Adaptation Model /experimental

INTERVENTIONS:
Behavioral: individualized nursing interventions based on the Roy Adaptation Model /experimental — The personal behaviors that could be related to recurrence (physiological, self-concept, role function, and mutual commitment) and the stimuli that caused recurrence (focal and affecting) were assessed, objectives were determined, and nursing interventions were carried out in line with these objectives. The interventions planned for diagnosing ineffective coping were selected according to the patients' needs among the "support coping" interventions under the title of the behavioral area in the Nursing Intervention Classification (NIC). A total of 10 individual interviews were made twice a week for about 45 to 60 minutes. The interviews were evaluated by determining the area specific Nursing outcome classification (NOC) (self respect, social support, mood management, role performance).
  Arms: experimental

SUMMARY:
Abstract Aim: This study aimed to determine the effect of individualized nursing interventions based on the Roy Adaptation Model on the recovery of alcohol addicts.

Method: This was an experimental study with pretest-posttest, follow-up, and a control group. It included 64 individuals who completed their detoxification process and met the inclusion criteria. The experimental group was provided with individualized care, and interventions were made in line with the Roy Adaptation Model. The personal behaviors that could be related to recurrence (physiological, self-concept, role function, and mutual commitment) and the stimuli that caused recurrence (focal and affecting) were assessed, objectives were determined, and nursing interventions were carried out in line with these objectives. The interventions planned for diagnosing ineffective coping were selected according to the patients' needs among the "support coping" interventions under the title of the behavioral area in the Nursing Intervention Classification (NIC).

The data were collected using an introductory information form, the Recovery Assessment Scale (RAS), the Turkish Version of the World Health Organization Quality of Life Instrument (WHOQOL-BREF-TR), and the Penn Alcohol Craving Scale (PACS).

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with alcohol use disorder according to DSM 5 Completed the detoxification phase were able to understand the scales and forms and maintain individual interviews were between 30 and 60 years of age

Exclusion Criteria:

* with a psychotic disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
The Recovery Assessment Scale (RAS) | A pretest was administered before starting the study and a posttest was administered 1 month later.
  The RAS was developed by Corrigan et al. (2004) and tested for validity and reliability in Turkish by Güler and Gürkan (2017). The scale consisted of 24 questions under 5 subscales. It was a five-point Likert type scale scored as follows: 1 = Strongly Disagree; 2 = Disagree; 3 = Not Sure; 4 = Agree; and 5 = Strongly Agree. The titles of the subscales were self-confidence and hope, seeking help, orientation to objectives and success, trust in the environment, and coping with the symptoms. Assessment could be made by scoring each item individually or over the total score. High total scores indicated high recovery. Cronbach's alpha coefficient of the Turkish form of the scale was 0.90.
World Health Organization Quality of Life Instrument | A pretest was administered before starting the study and a posttest was administered 1 month later.
  This health-related quality of life scale was developed by the World Health Organization and tested for validity and reliability in Turkish by Eser et al. The scale consisted of 27 questions that assessed individuals' physical, mental, social, and environmental well-being. Since each area independently represented the quality of life in its own domain, the area scores were calculated as between 4 and 20. High scores indicated a higher quality of life . The scale was selected by the substance addiction institute as the best scale that assessed the recovery of substance addiction. Cronbach's alpha coefficients of the subscales ranged between 0.73 and 0.84.
Penn Alcohol Craving Scale | A pretest was administered before starting the study and a posttest was administered after the study was completed. Follow-up testing was performed 1 month and 3 months after the end of the study.
  This was a five-item question form developed by Flannery et al. (1999) to assess the wish to drink alcohol (frequency, intensity, duration, resistance, and general craving). Each item was scored between 0 and 6. Thus, the maximum total severe craving score was 30. The scale was tested for validity and reliability in Turkish by Evren et al. (2008) with alcohol addicts, and its Cronbach alpha coefficient was found to be 0.94.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek AYAKDAŞ DAĞLI, Dr, Study Chair — İzmir Katip Çelebi Üniversity
Locations (1):
- İzmir Katip Çelebi University Ataturk Training and Research Hospital, Izmir, Karabağlar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No